CLINICAL TRIAL: NCT01774357
Title: Management and Detection of Atrial Tachyarrhythmias in Patients Implanted With BIOTRONIK DX Systems
Acronym: MATRIX
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA102
Record Dates: First submitted 2013-01-21; First posted 2013-01-24 (Estimated); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Atrial Fibrillation; Tachycardia; ICD Therapy; Thromboembolic Events; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia; Thromboembolism; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational registry study aiming to collect data on efficacy and safety of the single chamber Biotronik DX system with enhanced atrial diagnostics. The minimal follow-up period is 24 months. All analyses on the data will be done post-hoc; the study does not intend to confirm any pre-specified hypotheses.

DETAILED DESCRIPTION:
Enrollment (E0)

Timing:

• The enrollment (date of patient written informed consent) starts after implantation of a BIOTRONIK Lumax 540 VR-T DX ICD with Linoxsmart S DX or successor single chamber DX system according to current guidelines (primary or secondary prevention) but should not be later than 90 days after implantation.

Procedures:

* Check inclusion and exclusion criteria
* Patient information and written informed consent process
* Assignment of a unique study code
* ICD interrogation (re-programming if necessary)
* HMSC registration (recommended)
* Investigator assessment: appropriate atrial sensing

Documentation (note: where available the most recent assessment recorded within six months prior to hospital discharge shall be considered):

* Medical History:

  * Demographic data
  * General history of cardiovascular disease
  * Etiology of underlying heart disease
  * Cardiac events and symptoms
  * Documented supraventricular arrhythmia prior to implantation
* Device Interrogation

  * Date, home monitoring function, MRI scan
* AF history:

  * type (none, paroxysmal, persistent, permanent)
  * date of first diagnosis (if applicable)
  * EHRA classification (if applicable)
  * AF burden (if available)
  * CHA2DS2-VASc
  * Risk factors and comorbidities:
  * thyroid dysfunction
  * diabetes mellitus
  * COPD
  * sleep apnea
  * chronic renal disease
  * History of thromboembolic events or stroke
* Physical Examination:

  * Vital signs (SBP, DBP, height, body weight, BMI)
  * Current medication (substance class)
  * Heart failure indices
  * NYHA classification
  * BNP and NT-proBNP (only if determined in routine clinical practice)
  * LVEF (optional; echocardiography preferred, other methods accepted if no echo available)
  * ECG parameters (12 lead ECG; optional)
  * RR, PQ, and QT intervals
  * QRS width
  * rhythm disorders
  * clinical findings, morphology
* Implantation:

  * Indication (primary prevention, secondary prevention)
  * Type of procedure (first implantation / replacement)
  * RV lead:
  * Dislodgement / repositioning after implantation?
  * Sufficient amplitudes (Atrial; Ventricular) and thresholds (Ventricular)
  * Other clinical complications during / after implantation?
  * Final lead position at discharge (apical, septal, other)
  * Atrial dipole (with or without atrial wall contact at rest)
  * Ease of implantation as assessed by investigator
  * An extended questionnaire including more detailed information on implantation procedure, technique and initial measurements will be requested as an optional documentation where data are available

Follow-up Y1 and Y2

Timing:

• 12 and 24 months (+/-2 months) after enrollment respectively

Procedures:

* ICD interrogation / function check-up and re-programming if necessary
* Programmer download of all data not yet submitted to BIOTRONIK according to current working instruction
* Investigator assessment: appropriate atrial sensing

Documentation (note: where available the most recent assessment recorded between the current and the preceding visit shall be considered):

* Physical Examination:

  * Vital signs (SBP, DBP, height, body weight, BMI)
  * Current medication (substance class)
  * Heart Failure indices:
  * NYHA classification
  * BNP and NT-proBNP (only if determined in routine clinical practice)
  * LVEF (optional; echocardiography preferred, other methods accepted if no echo available)
  * ECG parameters (12 lead ECG; optional):
  * RR, PQ, and QT intervals
  * QRS width
  * rhythm disorders
  * clinical findings, morphology
* Device Interrogation

  * Date, home monitoring function, MRI scan

Event based documentation

* New-onset or worsening AF
* AF interventions
* Worsening heart failure
* Shock episode
* Thromboembolic events (CVA, TIA, PAE)
* Continuous surveillance / reporting of (serious) adverse events / (serious) adverse device effects

ELIGIBILITY:
Inclusion Criteria:

* Indication for implantation of a single chamber ICD (primary or secondary prevention) according to current guidelines
* Implanted with a BIOTRONIK Lumax 540 VR-T DX ICD with Linoxsmart S DX or successor single chamber DX system within 90 days prior to enrollment
* Written informed consent, willingness and ability to comply with the protocol

Exclusion Criteria:

* Age < 18 years
* Any limitation to contractual capability
* Female patients who are pregnant or breast feeding or plan a pregnancy during the course of the study
* Known active malignant disease or recovered from malignant disease within 2 years prior to enrollment
* Simultaneous participation in another study
* Life expectancy < 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for implantation of a single chamber ICD (primary or secondary prevention) according to current guidelines and after implantation of a BIOTRONIK Lumax 540 VR-T DX ICD with Linoxsmart S DX or successor single chamber DX system within 90 days prior to enrollment
Sampling Method: Probability Sample
Enrollment: 2054 (Actual)
Dates: Start 2013-01; Primary Completion 2018-09 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Frequency and types of AF-related complications | 24 months
Time to occurrence of first AF-related complication | 24 months
Time to AF-related intervention after detection of de novo or worsening AF | 24 months

SECONDARY OUTCOMES:
Frequency and type of complications related to implantation | 24 months
Frequency and type of lead-related complications | 24 months
All-cause mortality | 24 months
Cardiovascular hospitalization with days in hospital | 24 months
Significance of AF in acute decompensation of heart failure | 24 months
Interventions based on Home Monitoring information regarding AF | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, Prof. Dr., Principal Investigator — Herzzentrum Leipzig, Germany
Locations (1):
- Herzzentrum Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No